CLINICAL TRIAL: NCT00087295
Title: A Phase II Study of Depsipeptide (NSC-630176) In Patients With Advanced Transitional Cell Carcinoma Of The Urinary Tract Who Have Progressed After Receiving One Prior Chemotherapy Regimen For Advanced Disease
Brief Title: S0400, FR901228 in Treating Patients With Advanced Cancer of the Urothelium
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Permanently Closed Due to Poor Accrual
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000373886; U10CA032102 (NIH); S0400 (Other: SWOG)
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-10

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter; Urethral Cancer
Keywords: recurrent bladder cancer; stage IV bladder cancer; transitional cell carcinoma of the bladder; metastatic transitional cell cancer of the renal pelvis and ureter; recurrent transitional cell cancer of the renal pelvis and ureter; anterior urethral cancer; posterior urethral cancer; recurrent urethral cancer; urethral cancer associated with invasive bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Depsipeptides; romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Depsipeptide
  Interventions: Drug: Depsipeptide

INTERVENTIONS:
Drug: Depsipeptide — Depsipeptide wil be given 13 mg/m^2 through an intravenous (IV) over 4 hours on day 1, 8, and 15 for every 28 days (1 cycle = 28 days) until progression. Patients achieving a complete response (CR) will receive two additional cycles of treatment, and then be removed from protocol treatment.
  Other Names: FR901228; FK228

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as FR901228 (depsipeptide), work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well FR901228 works in treating patients with advanced cancer of the urothelium that has progressed or recurred after receiving one chemotherapy regimen.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response (confirmed complete and partial) in patients with advanced transitional cell carcinoma of the urothelium that has progressed after prior chemotherapy when treated with FR901228 (depsipeptide) .
* Determine progression-free and overall survival of patients treated with this drug.
* Determine the qualitative and quantitative toxic effects of this drug in these patients.
* Determine, preliminarily, the effects of this drug on reversing tumor promoter gene methylation in these patients.
* Correlate, preliminarily, tumor DNA in plasma with response or outcome in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive FR901228 (depsipeptide) IV over 4 hours on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response receive 2 additional courses of treatment.

Patients are followed every 3 months for 1 year and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed transitional cell carcinoma of the urothelium (bladder, renal pelvis, ureter, or urethra)

  * Metastatic disease

    * Node-positive, non-metastatic disease that is unresectable is allowed
  * Poorly differentiated transitional cell carcinoma OR predominant transitional cell carcinoma with rare foci of squamous differentiation or rare foci of adenocarcinoma allowed
* The following histologic types are not allowed:

  * Adenocarcinoma
  * Small cell carcinoma
  * Sarcoma
  * Squamous cell carcinoma
  * Mixed adeno/squamous/transitional histology
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 2 cm by conventional techniques OR ≥ 1 cm by spiral CT scan
  * Soft tissue disease irradiated within the past 2 months is not considered measurable
* Disease progression or recurrence after 1, and only 1, prior systemic chemotherapy regimen that included cisplatin or carboplatin for metastatic disease
* Not curable by surgery or radiotherapy
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* White blood cell (WBC) count ≥ 3,000/mm^3

Hepatic

* Aspartate aminotransferase (SGOT) / alanine aminotransferase (SGPT) ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin normal

Renal

* Creatinine ≤ 2 times ULN

Cardiovascular

* Corrected QT interval (QTc) < 500 msec
* Left ventricular ejection fraction (LVEF) > 40% by Multi Gated Acquisition Scan (MUGA)
* No New York Heart Association class III or IV congestive heart failure
* No myocardial infarction within the past year
* No uncontrolled dysrhythmias
* No poorly controlled angina
* No serious ventricular arrhythmia (ventricular tachycardia or ventricular fibrillation ≥ 3 beats in a row)
* No left ventricular hypertrophy on EKG
* No other significant cardiac disease

Other

* Potassium ≥ 4 mmol/L
* Magnesium ≥ 2 mg/dL
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No prior allergic reaction to compounds of similar chemical or biological composition to FR901228 (depsipeptide)
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy

Chemotherapy

* See Disease Characteristics
* At least 28 days since prior chemotherapy
* No prior FR901228 (depsipeptide)
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent hormonal therapy

Radiotherapy

* See Disease Characteristics
* More than 28 days since prior radiotherapy
* No concurrent radiotherapy

Surgery

* More than 28 days since prior surgery

Other

* Recovered from all prior therapy
* More than 28 days since prior intravesical therapy
* No concurrent hydrochlorothiazide
* No concurrent agent that causes QTc prolongation
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational histone deacetylase inhibitor agents or drugs (e.g., sodium valproate)
* No other concurrent anticancer therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2004-06; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Probability of response (confirmed complete and partial) | From date of registration to progression or death from any cause, whichever came first, assessed up to 3 years

SECONDARY OUTCOMES:
Progression-free survival | From date of registration to progression or death from any cause, whichever came first, assessed up to 3 years
Overall survival | From date of registration to progression or death from any cause, whichever came first, assessed up to 3 years
Number and grade of adverse events | From date of registration to progression or death from any cause, whichever came first, assessed up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Daniel P. Petrylak, MD, Study Chair — Herbert Irving Comprehensive Cancer Center